CLINICAL TRIAL: NCT00619151
Title: A Randomized Study to Compare Sizing, Implant Techniques, & Hemodynamic Performance Between the CarboMedics Supra-annular Top Hat Valve and the St. Jude Medical Regent Valve in the Aortic Position.
Brief Title: CarboMedics Top Hat vs St. Jude Medical Regent Valve Comparing Sizing and Hemodynamics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to lack of elegible patient enrollment
Sponsor: Sorin Group USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RVSS-1H
Record Dates: First submitted 2008-01-10; First posted 2008-02-20 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-09

CONDITIONS: Aortic Valve Disease
Keywords: aortic valve; heart valve; valve replacement; Valve disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CarboMedics Supra-annular Top Hat Valve
  Interventions: Device: Top Hat
- 2 (Active Comparator): St. Jude Medical Regent Valve
  Interventions: Device: Regent

INTERVENTIONS:
Device: Top Hat — Implant of CarboMedics Top Hat mechanical valve.
  Arms: 1
Device: Regent — Implant of the St. Jude Medical Regent mechanical valve
  Arms: 2

SUMMARY:
The purpose of this study is to compare the sizing and implant techniques between the CarboMedics Top Hat supra-annular valve and the St. Jude Medical Regent valve.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are indicated for implant with a mechanical valve prosthesis in the aortic position according to the current practice for valve selection at the center.

Exclusion Criteria:

* Patients < 18 years of age
* Emergency surgery
* Pre-existing valve prosthesis
* Aortic root replacement
* Active endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Top Hat Valve: CarboMedics Supra-annular Top Hat Valve
- St.Jude Valve: St. Jude Medical Regent Valve
Period: Overall Study
Arm/Group | Top Hat Valve | St.Jude Valve
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Study terminated prior to followup | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Top Hat Valve | St.Jude Valve | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Customized [Number; unit: participants]
  <18 years | 0 |  | 0
  >= 18 years | 2 |  | 2
Sex/Gender, Customized [Number; unit: participants]
  Unknown | 2 |  | 2
  Female | NA — Previous values entered in error. Study records archived and not accessible. |  |
  Male | NA — Study records archived and not accessible. |  |
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Effective Orifice Area (EOA)
Description: Effective Orifice Area of the prosthetic valve measured via echocardiography to determine physiological area of blood flow through the valve.
Time Frame: 6 month evaluation
Population: Analysis not performed due to study termination prior to analysis period.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Top Hat Valve | St.Jude Valve
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Aortic Mean Gradient
Description: Mean gradient measured across the aortic prosthetic valve via echocardiography to determine mean pressure of blood flow across the valve.
Time Frame: 6 months
Population: Analysis not performed due to study termination prior to analysis period.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Top Hat Valve | St.Jude Valve
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of hospital stay after surgery, an average of 4 days.
Description: Adverse event information collected during hospital stay
Arm/Group | Top Hat Valve | St.Jude Valve
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to low enrollment resulted in only 2 patients. Insufficient data for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less